CLINICAL TRIAL: NCT00317252
Title: Angiotensin Converting Enzyme Inhibitors and Contrast Induced Nephropathy in Patients Receiving a Cardiac Catheterization "The CAPTAIN Trial"
Brief Title: Angiotensin Converting Enzyme Inhibitors & Contrast Induced Nephropathy in Patients Receiving a Cardiac Catheterization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Dr. Shamir Mehta, Associate Professor of Medicine, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-005
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Failure
Keywords: contrast induced nephropathy; contrast nephropathy; contrast media; kidney diseases; angiotensin converting enzyme inhibitors
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hold ACEI or ARB (Experimental): Angiotensin converting enzyme inhibitor or angiotensin receptor blocker held >= 24 hours pre-cardiac catheterization and restarted post-catheterization after creatinine measurement (48-96 hours post)
  Interventions: Drug: Hold ACEI or ARB
- Continue ACE1 or ARB (Other): Randomized to continue on prescribed ACE1 or ARB
  Interventions: Drug: Hold ACEI or ARB

INTERVENTIONS:
Drug: Hold ACEI or ARB — Angiotensin converting enzyme inhibitor or angiotensin receptor blocker held at least 24 hours pre-cardiac catheterization and restarted 48-96 hours post-catheterization (after creatinine measurement)
  Other Names: Includes all ACE inhibitors or ARBs

SUMMARY:
The purpose of this study is to determine if patients should stop taking their angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) around the time of their angiogram in order to prevent contrast induced nephropathy (CIN).

DETAILED DESCRIPTION:
There are approximately 4000 coronary angiograms performed annually at the Hamilton General Hospital to diagnose and treat coronary artery disease. Many of the patients undergoing this procedure have mild kidney disease. Exposure to the contrast dye used in the procedure puts them at risk of worsening kidney function, a condition called contrast induced nephropathy (CIN) which is associated with significant morbidity and mortality. Many of these patients are also on an antihypertensive drug called an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB). Their effects on the kidney during contrast exposure are not known. Our understanding of how the drug works leads us to believe that the use of these drugs around the time of contrast exposure may have detrimental effects on the kidney.

The purpose of this study is to determine if patients should continue taking or stop taking their ACE inhibitor or ARB around the time of their angiogram in order to prevent CIN.

Patients undergoing an elective coronary angiogram with mild kidney disease and currently taking an ACE inhibitor or ARB will be randomly divided into two groups. One group will continue taking their ACE inhibitor or ARB while the other group will stop taking their ACE inhibitor or ARB for at least 24 hours before and will resume their ACE inhibitor or ARB 48 to 96 hours after their angiogram. In both groups, kidney function will be assessed by means of a simple blood test both before and 48 to 96 hours after the angiogram. By doing this, we can determine which group had more kidney damage and which group had less kidney damage from the contrast exposure. We suspect that patients who do not take their ACE inhibitor around the time of their angiogram will have less kidney damage. All patients will receive the accepted measures for preventing kidney disease from contrast dye exposure.

CIN is associated with significant morbidity and mortality. If the use of ACEIs during coronary angiograms are associated with an increased risk of CIN, then these patients may benefit from holding their ACEI around the time of their procedure potentially improving their outcomes. This is a low cost intervention that could potentially change practice, reduce morbidity, save lives and pave the way for larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Angiography in >= 24hrs from enrolment
* Documented Cr >= 150 within 3 months before cardiac catheterization AND/OR documented Cr >= 132umol/L within 1 week Before Cardiac Catheterization
* Currently Taking an ACE Inhibitor

Exclusion Criteria:

* Patients with end stage renal disease (for example, patient on dialysis)
* Emergency Cardiac Catheterization with insufficient time to hold the ACEI
* Acute Pulmonary Edema

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy (creatinine rise of 44umol/L or 25% compared to the pre-randomization creatinine level) at 48-96hrs | 48 - 96 hours post-cardiac catheterization

SECONDARY OUTCOMES:
Change in serum creatinine at 48-96hrs | 48 - 96 hours post-cardiac catheterization
Change in creatinine clearance at 48-96hrs | 48 - 96 hours post-cardiac catheterization
Death, Myocardial Infarction, Stroke, Congestive Heart Failure, dialysis, major bleeding, minor bleeding, hypertension, re-hospitalization at 48-96hrs. | 48 - 96 hours post-cardiac catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Shamir R Mehta, MD MSc, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Bainey KR, Rahim S, Etherington K, Rokoss ML, Natarajan MK, Velianou JL, Brons S, Mehta SR; CAPTAIN Investigators. Effects of withdrawing vs continuing renin-angiotensin blockers on incidence of acute kidney injury in patients with renal insufficiency undergoing cardiac catheterization: Results from the Angiotensin Converting Enzyme Inhibitor/Angiotensin Receptor Blocker and Contrast Induced Nephropathy in Patients Receiving Cardiac Catheterization (CAPTAIN) trial. Am Heart J. 2015 Jul;170(1):110-6. doi: 10.1016/j.ahj.2015.04.019. Epub 2015 Apr 18. PMID 26093871